CLINICAL TRIAL: NCT02669888
Title: Efficacy and Safety of Topical Indigo Naturalis in Treating Atopic Dermatitis: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Indigo Naturalis in Treating Atopic Dermatitis Topically
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MOST 104-2325-B-182A-005
Record Dates: First submitted 2015-12-28; First posted 2016-02-01 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Atopic Dermatitis
Keywords: Indigo Naturalis; Atopic Dermatitis; TCM
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Qingdai compound

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Indigo naturalis ointment (Experimental): 1. Form: ointment
  2. Dose: each gram of ointment contains 200µg of indirubin
  3. Dosing schedule: apply 0.5g of ointment per 10 x 10 dermatitis lesion twice daily
  Interventions: Drug: Indigo naturalis ointment
- Placebo (Placebo Comparator): 1. Form: ointment
  2. Dose: vehicle
  3. Dosing schedule: apply 0.5g of ointment per 10 x 10 dermatitis lesion twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Indigo naturalis ointment — Every 10 x 10 cm area of lesion requires 0.5 g of ointment, applied twice daily (morning and evening, separated by approximately 12±2 hours) for 6 weeks.
  Other Names: Lindioil ointment
  Arms: Indigo naturalis ointment
Drug: Placebo — Every 10 x 10 cm area of lesion requires 0.5 g of ointment, applied twice daily (morning and evening, separated by approximately 12±2 hours) for 6 weeks.
  Arms: Placebo

SUMMARY:
Atopic dermatitis (AD) is a chronic inflammatory skin disorder that most commonly occurs in children. The aims of this project are:

1. To evaluate the efficacy of indigo naturalis ointment in treating AD topically;
2. To evaluate the safety of indigo naturalis ointment in treating AD topically;
3. To investigate whether indigo naturalis ointment treatment is associated with a change in total IgE, cytokines, eosinophils, and CRP in patients with AD;
4. To evaluate whether indigo naturalis ointment treatment improves the quality of life in patients with AD.

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is a chronic inflammatory skin disorder that most commonly occurs in children. AD is characterized by itchy and dry skin that affects approximately 5 to 20% of children in the world. Currently, corticosteroids are the most widely prescribed medication in treating AD; however, there are concerns regarding the side effects such as skin atrophy, telangiectasia, striae, folliculitis and adrenocortical suppression that inhibits growth in children. Many patients and families seek complementary and alternative medications such as traditional Chinese medicine (TCM). In TCM, indigo naturalis has been used to treat various infectious and inflammatory skin diseases for hundreds of years. Ancient TCM literature has recorded that indigo naturalis is also effective in treating facial eczema (AD) in infants.

The aims of this project are: (1) To evaluate the efficacy of indigo naturalis ointment in treating AD topically; (2) To evaluate the safety of indigo naturalis ointment in treating AD topically; (3) To investigate whether indigo naturalis ointment treatment is associated with a change in total IgE, cytokines, eosinophils, and CRP in patients with AD; (4) To evaluate whether indigo naturalis ointment treatment improves the quality of life in patients with AD.

ELIGIBILITY:
Inclusion Criteria:

1. Between 6 and 65 years old, female or male.
2. Atopic dermatitis fulfilling the diagnostic criteria of Williams et al.
3. Atopic dermatitis involving <40% of BSA. (Base on the BSA result of Screening)
4. An Investigator's Global Assessment (IGA) score of 2, 3 or 4 which corresponds to mild, moderate or severe disease. (Base on the IGA result of Screening)
5. Female patients of child-bearing age with negative pregnancy test at screening.
6. Female patients of child-bearing age that agree to continue using birth control measures approved by the investigator and agree not to lactate for the duration of the study.
7. Agree to only receive stable doses of an additive-free, basic bland emollient for at least 7 days before baseline (day0)
8. Willing to comply with study protocol and agree to sign an informed consent form.

Exclusion Criteria:

1. Having a history of topical or systematical hypersensitivity to indigo naturalis or its excipient (e.g. beeswax) in ointment
2. Undergoing phototherapy (e.g. UVB, PUVA) or systemic therapy (e.g. Immunosuppressive agents) within 30 days.
3. Having used topical therapy (e.g. topical corticosteroids) for dermatitis within 7 days before the first application of the study medication.
4. Having a significant concurrent disease, such as: significant abnormalities in hematology, severe uncontrolled metabolic syndrome (e.g., hypertension, diabetes mellitus, metabolic arthritis, hyperthyroidism), psychiatric disease, cancer or AIDS.
5. Having abnormal liver or renal function (AST/ALT >3 x ULN, creatinine >2.0 mg/dl).
6. Women who are lactating, pregnant or preparing to be pregnant.

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Percentage change in Eczema Area Severity Index (EASI) scores from baseline to week 6 | 6 weeks
  The Eczema Area and Severity Index (EASI) is used to measure the disease severity of erythema, infiltration/papulation, excoriation, and lichenification each on a scale of 0 to 3 (none to severe) as well as the percentage of disease area on a scale of 0 to 6 for the head ⁄ neck, upper limb, trunk and lower limb body regions. Each body region score is calculated by multiplying the disease severity score by the disease area score and by the multiplier. The scores are summed to give the total EASI score, ranging from 0 to a maximum 72.
  The mean percentage change in EASI = (EASI baseline-EASI post-treat) / EASI baseline x 100%

SECONDARY OUTCOMES:
Proportion of subjects who have achieved EASI-50, EASI-75, and EASI-90 after 6 weeks of treatment | 6 weeks
  It is defined as at least 50%, 75%, and 90% reduction in EASI score relative to the baseline.
Proportion of subjects with a change in Investigator's Global Assessment (IGA, range 0-5) from baseline to week 6. | 6 weeks
  1. Proportion of subjects with an IGA score of 0 (clear) or 1 (almost clear) at week 6.
  2. Proportion of subjects with ≥ 2 point improvement in IGA at week 6.
The mean percentage change in Total Body Surface Area involved with AD (BSA, range 0%-100%) from baseline to week 6. | 6 weeks
  BSA is total Body Surface Area involved, ranging from 0% (none) to 100% (total body surface involved)
The mean change in pruritus score (10-cm visual analogue scale) from baseline to week 6. | 6 weeks
  Visual Analogue Scale (VAS) for pruritus severity rates from 0 (no itching) to 10 (very severe itching)
Clinical-immunological correlation between the treatment outcome and the changes in the level of immunoglobin E (IgE), cytokines, eosinophil count, and C-reactive protein (CRP) in the peripheral blood from baseline to week 6. | 6 weeks
  Measuring the correlations of treatment by EASI score and BSA, with the changes in IgE, eosinophils, cytokines (IL-1β, IL-6, TNF-α…) from baseline to week 6.
The mean change in Dermatology Life Quality Index (DLQI)from baseline to week 6 | 6 weeks
  The DLQI is a self-administered 10-item questionnaire, ranges from 0 (best) to 30 (worst); the higher the score, the more quality of life is impaired.
  For subjects from age 6 to age 16, children's DLQI (CDLQI) will used.
Physician's Global Assessment (PGA ) at week 6. | 6 weeks
  0 = Symptoms cleared or excellent improvement of 90-100%; 1 = Marked improvement of 75-89%; 2 = Moderate improvement of 50-74%; 3 = Slight improvement of 3049%; 4 = No appreciable improvement of 029%; 5 = Worsening of the condition
Subject's Global Assessment (SGA) at week 6. | 6 weeks
  0 = Symptoms cleared or excellent improvement of 90-100%; 1 = Marked improvement of 75-89%; 2 = Moderate improvement of 50-74%; 3 = Slight improvement of 3049%; 4 = No appreciable improvement of 029%; 5 = Worsening of the condition

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Ku Lin, MD., PhD., Principal Investigator — Chang Gung Memorial Hospital
Locations (3):
- Taiwan (3):
  - Chang Gung Memorial Hospital at Keelung, Kelung, Taiwan
  - Chang Gung Memorial Hospital at Taipei, Taipei, Taiwan
  - Chang Gung Memorial Hospital at Linkou, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin YK, Chang SH, Yang CY, See LC, Lee BH, Shih IH. Efficacy and safety of indigo naturalis ointment in Treating Atopic Dermatitis: A randomized clinical trial. J Ethnopharmacol. 2020 Mar 25;250:112477. doi: 10.1016/j.jep.2019.112477. Epub 2019 Dec 12. PMID 31838180